CLINICAL TRIAL: NCT07267468
Title: Effectiveness of an mHealth Intervention, Based on Rehabilitation and a Personalised Nutrition Plan, in the Recovery and Improvement of Dysphagia in Patients Diagnosed With Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Collaborators: Andalusian Health Service (Other Government)
Responsible Party: Principal Investigator, Antonio Jesús Marín Paz, Collaborator Investigator, University of Cadiz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP-0331-2022-C3-F2
Record Dates: First submitted 2025-11-13; First posted 2025-12-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Stroke; Deglutition Disorders
Keywords: Stroke; Deglutition Disorders; Pneumonia, Aspiration; Nutrition; Rehabilitation; mHealth
MeSH Terms: conditions — Stroke; Deglutition Disorders; Pneumonia, Aspiration

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The random allocation of participants will also be blinded to the researchers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth Group (Experimental): This group will receive the mHealth intervention via the mobile application "DegluApp".
  Interventions: Other: mHealth intervention
- No intervention Group (No Intervention): This group will perform conventional care according to the healthcare centers' protocols.

INTERVENTIONS:
Other: mHealth intervention — The intervention consists of using the validated mobile application "DegluApp", which contains recommendations and exercises related to nutrition, physical activity, rehabilitation, warning signs, and games pertinent to the daily life of a person with post-stroke dysphagia.
  Arms: mHealth Group

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of an mHealth intervention as a complement to usual clinical practice for the improvement and recovery of dysphagia in patients who have suffered a stroke. The main question it aims to answer is:

- Does the mHealth intervention improve the recovery of dysphagia in post-stroke patients compared to usual care alone?

Researchers will compare patients receiving the mHealth intervention plus usual care to see if the combined approach leads to better dysphagia outcomes, reduced negative consequences (e.g., malnutrition, pneumonia), and improved quality of life compared to usual care alone.

Participants will be recruited and:

* Receive a diagnosis and usual care for post-stroke dysphagia.
* Be assigned to either the mHealth intervention group (using a smartphone/tablet app for information and follow-up) or the control group (usual care only).
* Be followed up to assess dysphagia recovery, reduction in negative outcomes (like aspiration pneumonia, dehydration), and changes in quality of life.

DETAILED DESCRIPTION:
Stroke is one of the leading causes of death and disability globally, and is associated with negative complications and increased socio-health costs. Among the complications derived from a stroke is dysphagia, defined as difficulty swallowing, which is associated with increased morbidity and mortality. Up to 80% of patients who have a stroke have difficulty swallowing. Furthermore, this is more pronounced in older adults, as the oropharyngeal swallowing response is affected in this population. Dysphagia is a significant predictor of negative outcomes such as malnutrition, dehydration, tracheobronchial aspiration, pneumonia, and death derived from pneumonia, low mood, and depression, etc. These consequences reduce the perception of quality of life for patients with dysphagia. Early intervention and the continuity of this intervention at home reduce the negative consequences of dysphagia. Currently, the majority of the population owns a smartphone or tablet and uses mobile applications (apps) in their daily lives to communicate, seek information, etc. Mobile technology can be a useful support tool for health professionals, facilitating information and follow-up for post-stroke patients with dysphagia and empowering patients and family members in managing their health. The general objective of this study is to evaluate the efficacy of an mHealth intervention, as a complement to usual clinical practice, for the improvement and recovery of dysphagia in patients who have suffered a stroke.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years or older.
* Patients with any degree of impairment in swallowing/oropharyngeal dysphagia to liquids following a stroke (ACV).

Exclusion Criteria:

* Hospitalized patients presenting any type of visual barrier.
* Patients in terminal palliative care.
* Patients in the final days of life phase.
* Patients with severe cognitive impairment.
* Patients with a language barrier regarding the use of the App.

Subject Withdrawal Criteria:

* Revocation of consent. In this case, the subject will exit the study and will not be replaced by another subject, being considered a "loss".
* Lack of adherence to the prescribed training plan exceeding 20% of the scheduled sessions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2026-01-30 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Dysphagia Improvement and Recovery | Day 1, 3 months, 6 months, and 9 months
  Dysphagia Improvement and Recovery. Dichotomous qualitative variable: Yes, No.
Type of texture | Day 1, 3 months, 6 months, and 9 months
  Type of texture and volume the patient follows in their habitual diet. Categorical qualitative variable: Liquid, Nectar, Honey, Pudding.
Volume allowed when swallowing | Day 1, 3 months, 6 months, and 9 months
  Volume the patient follows in their habitual diet. Categorical qualitative variable: 5 mL, 10 mL, and 20 mL
Acceptable viscosity when swallowing | Day 1, 3 months, 6 months, and 9 months
  Measured using the Volume-Viscosity Swallow Test (V-VST). The test is performed using three different viscosities (thin liquid, nectar-thick, and pudding-thick) and three different volumes 3 ml, 5 ml, and 20 ml) to determine the volume-viscosity combination that is safest and most efficient for the patient. It is a clinical diagnostic tool used to evaluate the efficacy and safety of a patient's swallowing function (deglutition) by systematically challenging it with a controlled set of liquid volumes and viscosities. It contains two main safety and efficiency markers. For the Safety Scale (aspiration/penetration), levels typically range from a minimum of 0 (no safety issues detected) to a maximum of 2 (indicating severe issues like persistent cough or desaturation). Similarly, the Efficiency Scale might range from Level 0 (efficient swallow) to Level 1 (reduced efficiency).

SECONDARY OUTCOMES:
Perceived quality of life | Day 1, 3 months, 6 months, and 9 months
  Categorical qualitative variable: EuroQoL 5 Dimensions - 5 Levels (EuroQoL 5D-5L). They are scored using a 5-point Likert scale (1. No problem; 5. Unable). The sixth dimension scores ranging from 0 (worst health status) to 100 (best health status).
Weight | Day 1, 3 months, 6 months, and 9 months
  Continuous quantitative variable: kg.
Height | Day 1, 3 months, 6 months, and 9 months
  Continuous quantitative variable: cm.
Body Mass Index | Day 1, 3 months, 6 months, and 9 months
  Continuous quantitative variable: kg/m².
Anthropometric variables | Day 1, 3 months, 6 months, and 9 months
  Circumferences (arm and calf). Continuous quantitative variable. Unit of measurement: Millimeters (mm).
Dynamometry | Day 1, 3 months, 6 months, and 9 months
  Body dynamometry measures the maximum voluntary isometric contraction (MVIC), which is the greatest force a muscle can generate without changing its length, or isokinetic strength, which is the force generated across a range of motion at a constant angular velocity. The primary variable is force, which reflects the muscle's ability to produce tension. Continuous quantitative variable. In general clinical practice using a handgrip dynamometer (a common and standardized measure), minimum values can be very low (e.g., under 10 kg for older, frail, or sarcopenic individuals). Very low values are often indicative of frailty or severe muscle wasting. Maximum values can reach or exceed 60 kg for strong, healthy, and athletic adult men.
  Unit of measurement: kg.
Diet | Day 1, 3 months, 6 months, and 9 months
  Diet serves to classify subjects into distinct, non-ordered categories based on their primary eating patterns (omnivore, vegetarian, vegan, pescatarian, keto, mediterranean). Nominal qualitative variable.
Dietary Intake | Day 1, 3 months, 6 months, and 9 months
  Categorical qualitative variable: 25%, 50%, 75%, and 100%.
Sarcopenia | Day 1, 3 months, 6 months, and 9 months
  Dichotomous qualitative variable: SARC-F Questionnaire (Strength, Assistance in walking, Rise from a chair, Climb stairs, Falls). The SARC-F measures five key components related to muscle function and strength, which are reported by the individual being assessed. Each component is scored from 0 to 2 points. The total score is the sum of the points from the five components, resulting in a range from a minimum value of 0, which indicates the lowest risk for sarcopenia, to a maximum value of 10 (5 components x 2 points/component), which indicates the highest risk for sarcopenia. The SARC-F is primarily interpreted using a simple cut-off point for screening: a score of >4 points is considered positive and indicates a high risk for sarcopenia.
Nutritional Status | Day 1, 3 months, 6 months, and 9 months
  Discrete quantitative variable: Mini-Nutritional Assessment (MNA). It is designed to identify elderly individuals who are malnourished or at risk of malnutrition. It comprehensively evaluates several factors that influence nutritional status, including anthropometric measurements, general lifestyle and functional capacity, dietary changes, and self-perception of health and nutritional status. It is crucial for early intervention in geriatric care. The MNA produces a single score ranging from a minimum value of 0 (indicating severe malnutrition) to a maximum value of 30 (indicating satisfactory nutritional status). Scores are then grouped into categories: <17 (malnourished), 17.5 to 23.5 (at risk of malnutrition), and > 24 (well-nourished).
Caregiver Burden | Day 1, 3 months, 6 months, and 9 months
  Categorical qualitative variable: Zarit Burden Interview (ZBI). The ZBI assesses the subjective stress, strain, and emotional distress felt by the caregiver. It consists of 22 items (in the full version) rated on a 5-point Likert scale ranging from 0 (Never) to 4 (Nearly always). The total score is the sum of the points from all 22 items, resulting in a range from a minimum value of 0, which indicates no burden is perceived by the caregiver, to a maximum value of 88 (22 items x 4 points/item), which indicates the highest level of perceived burden. The score is interpreted using established cut-off points to categorize the level of burden: scores typically ranging from 0 to 20 suggest no or minimal burden; scores between 21 and 40 indicate mild to moderate burden; scores from 41 to 60 suggest moderate to severe burden; and scores from 61 to 88 denote severe burden.
Caregiver Strain | Day 1, 3 months, 6 months, and 9 months
  Discrete quantitative variable: Caregiver Strain Index. The CSI measures the caregiver's perception of strain across three main domains related to their caregiving role: Financial Strain, Physical Strain, and Emotional and Social Strain. The questionnaire consists of ten statements about common sources of strain. The caregiver responds to each item with a simple "yes" (strain is present) or "no" (strain is absent). The total score is calculated by summing the number of "yes" responses. The score ranges from a minimum value of 0, which indicates no strain is perceived by the caregiver, to a maximum value of 10 (10 items x 1 point/item), which indicates the highest level of perceived strain. The CSI is interpreted using a key cut-off point: a score of >7 points is generally considered clinically significant, indicating a high level of caregiver strain.
Fat Mass | Day 1, 3 months, 6 months, and 9 months
  The total amount of stored fat in the body, including essential (vital for life and reproductive functions) and non-essential (storage) fat. It's a key component in assessing body composition, often used to determine the degree of obesity and related health risks. Continuous quantitative variable.
  A healthy minimum body fat percentage for men is around 5%, and for women, around 10-13% (due to essential fat). Absolute minimum for survival is closer to 1-3% for men and 8-12% for women, but these are dangerously low values. Maximum value can exceed 50% of total body weight in cases of severe obesity. There is no biological maximum, but values over 40% often indicate high health risk.
  Unit of measurement: Kilograms (kg or %).
Fat-Free Mass | Day 1, 3 months, 6 months, and 9 months
  The portion of the body that does not contain fat. It is composed primarily of muscle, bone, water, and internal organs (e.g., bone mineral mass, protein mass). It represents the metabolically active tissue and is a major determinant of Basal Metabolic Rate (BMR). Continuous quantitative variable. Minimum value varies widely based on height and body type, but generally represents a large proportion of total weight, typically over 50% of total body mass. Maximum value highly dependent on the individual's size, muscle mass, and hydration status. Unit of measurement: Kilograms (kg).
Body Water | Day 1, 3 months, 6 months, and 9 months
  The total amount of water in the human body, encompassing both Intracellular Fluid (ICF) and Extracellular Fluid (ECF). Water is the largest component of Fat-Free Mass and is essential for nearly all physiological functions. It is a key indicator of hydration status. Continuous quantitative variable. Minimum value represents a large part of the body. Healthy adult men typically have 50-65% of their body mass as water, while healthy adult women typically have 45-60%. Values below this can indicate severe dehydration. Maximum value cannot biologically exceed the physiological upper limit (around 65-70% for the general population), as body water is homeostatically controlled. Excessively high values may indicate conditions like edema. Unit of measurement: Liters (L), Kilograms (kg), or Percentage (%) of total body weight.
Phase Angle | Day 1, 3 months, 6 months, and 9 months
  A raw measure derived from Bioelectrical Impedance Analysis (BIA) that relates the resistance and reactance of body tissues. It is a non-invasive indicator of cellular health, integrity, and function. A higher phase angle is generally associated with greater cell membrane integrity, better nutritional status, and greater muscle mass. A lower angle may indicate cell breakdown, poor health, or malnutrition. Minimum value can be as low as 2º or 3º in severely malnourished, ill, or elderly patients. Maximum value typically ranges up to 9º or 10º in healthy, muscular, or athletic individuals. Unit of measurement: Degrees (º).

OTHER OUTCOMES:
Sex | Day 1
  Dichotomous qualitative variable: Female, Male.
Age | Day 1
  Discrete quantitative variable: years.
Presence of caregiver | Day 1
  Dichotomous qualitative variable: Yes, No.
Degree of dependence for performing Activities of Daily Living | Day 1, 3 months, 6 months, and 9 months
  Categorical qualitative variable: Barthel Index. It is a foundational ordinal scale used primarily in rehabilitation and geriatric medicine to measure a person's level of independence in activities of daily living (ADLs) and functional mobility. It assesses ten essential areas: feeding, bathing, grooming, dressing, bowel control, bladder control, toilet use, transfers (bed to chair), mobility (walking or wheelchair), and climbing stairs. The total score reflects the individual's ability to perform these tasks with or without assistance, providing a clear indication of their care needs and the effectiveness of rehabilitation interventions. The Barthel Index ranges from a minimum value of 0, which signifies a totally dependent state requiring maximum assistance in all activities, to a maximum value of 100, which indicates complete independence in all ten functional areas.
Frailty | Day 1, 3 months, 6 months, and 9 months
  Through Fried criteria. It is a widely recognized and simple clinical method used to identify and classify the physical frailty status of older adults. It specifically focuses on the physical decline associated with aging. The result of the Fried Criteria is a count of the deficits (criteria) met, ranging from 0 to 5. Minimum value: 0, which indicates the individual is considered Non-frail (or Robust). Maximum value: 5, which means the individual meets all five criteria, indicating Severe Frailty. The results are typically categorized into three clinical states: Robust/Non-frail (0 criteria met), Pre-frail (1 or 2 criteria met), Frail (3 or more criteria met).
Risk of falls | Day 1, 3 months, 6 months, and 9 months
  Categorical qualitative variable: Falls Risk Detection Scale. It is a clinical screening tool used primarily in hospital and institutional settings to assess a patient's risk of falling. Its main purpose is to quickly identify individuals who require preventative measures to reduce their risk of falls during their stay. Minimum value: 0, indicating the lowest risk of falling. Maximum value: The maximum possible score can vary significantly, often up to 90 or more, indicating the highest risk of falling. Score Range: Low risk (0-24 points), moderate risk (25-50 points), high risk (>50 points).
Hospital admissions | Day 1, 3 months, 6 months, and 9 months
  Discrete quantitative variable: number of admissions.
Length of time a patient remains in the hospital | Day 1, 3 months, 6 months, and 9 months
  Continuous quantitative variable: days.
Economic cost | Day 1, 3 months, 6 months, and 9 months
  Continuous quantitative variable: euros. Will be calculated by multiplying the days of admission or hospital stay by the daily cost of life.
Presence of aspiration | Day 1, 3 months, 6 months, and 9 months
  Discrete quantitative variable: number of aspiration episodes.
Presence of respiratory infection | Day 1, 3 months, 6 months, and 9 months
  Discrete quantitative variable: number of respiratory infection episodes.
Presence of aspiration-derived pneumonia | Day 1, 3 months, 6 months, and 9 months
  Discrete quantitative variable: number of aspiration-derived pneumonia episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Sánchez-Sánchez, Ph.D., Principal Investigator — University of Cadiz. Andalusian Healthcare Service
Locations (1):
- Faculty of Nursing. Punta Europa University Hospital, Algeciras, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data obtained in the study will be anonymized and will be published collectively in a database at the time of the publication of the research results.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study Protocol: October 2025. Informed Consent Form: October-November 2025. Statistical Analysis Plan: October-November 2025. Database of results: At the time of the publication of the research results.
Access Criteria: All data will be incorporated in open access both into this research protocol and at the time of the publication of the research results.

REFERENCES:
- [Background] Hernandez G, Garin O, Dima AL, Pont A, Marti Pastor M, Alonso J, Van Ganse E, Laforest L, de Bruin M, Mayoral K, Serra-Sutton V, Ferrer M; ASTRO-LAB Group. EuroQol (EQ-5D-5L) Validity in Assessing the Quality of Life in Adults With Asthma: Cross-Sectional Study. J Med Internet Res. 2019 Jan 23;21(1):e10178. doi: 10.2196/10178. PMID 30672744
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Background] Lim ML, Yong BYP, Mar MQM, Ang SY, Chan MM, Lam M, Chong NCJ, Lopez V. Caring for patients on home enteral nutrition: Reported complications by home carers and perspectives of community nurses. J Clin Nurs. 2018 Jul;27(13-14):2825-2835. doi: 10.1111/jocn.14347. Epub 2018 Apr 22. PMID 29518266
- [Background] Vellas B, Guigoz Y, Garry PJ, Nourhashemi F, Bennahum D, Lauque S, Albarede JL. The Mini Nutritional Assessment (MNA) and its use in grading the nutritional state of elderly patients. Nutrition. 1999 Feb;15(2):116-22. doi: 10.1016/s0899-9007(98)00171-3. PMID 9990575
- [Background] Sanchez-Rodriguez D, Marco E, Davalos-Yerovi V, Lopez-Escobar J, Messaggi-Sartor M, Barrera C, Ronquillo-Moreno N, Vazquez-Ibar O, Calle A, Inzitari M, Piotrowicz K, Duran X, Escalada F, Muniesa JM, Duarte E. Translation and Validation of the Spanish Version of the SARC-F Questionnaire to Assess Sarcopenia in Older People. J Nutr Health Aging. 2019;23(6):518-524. doi: 10.1007/s12603-019-1204-z. PMID 31233072
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Guillen-Sola A, Marco E, Martinez-Orfila J, Donaire Mejias MF, Depolo Passalacqua M, Duarte E, Escalada F. Usefulness of the volume-viscosity swallow test for screening dysphagia in subacute stroke patients in rehabilitation income. NeuroRehabilitation. 2013;33(4):631-8. doi: 10.3233/NRE-130997. PMID 24018371
- [Background] Ortega-Martin ME, Lucena-Anton D, Luque-Moreno C, Heredia-Rizo AM, Moral-Munoz JA. [Commercial mobile applications in the therapeutic approach to stroke: Review in main application repositories and scientific evidence]. Rev Esp Salud Publica. 2019 Jun 12;93:e201906035. Spanish. PMID 31204385
- [Background] Teasell R, Salbach NM, Foley N, Mountain A, Cameron JI, Jong A, Acerra NE, Bastasi D, Carter SL, Fung J, Halabi ML, Iruthayarajah J, Harris J, Kim E, Noland A, Pooyania S, Rochette A, Stack BD, Symcox E, Timpson D, Varghese S, Verrilli S, Gubitz G, Casaubon LK, Dowlatshahi D, Lindsay MP. Canadian Stroke Best Practice Recommendations: Rehabilitation, Recovery, and Community Participation following Stroke. Part One: Rehabilitation and Recovery Following Stroke; 6th Edition Update 2019. Int J Stroke. 2020 Oct;15(7):763-788. doi: 10.1177/1747493019897843. Epub 2020 Jan 27. PMID 31983296
- [Background] Marin S, Serra-Prat M, Ortega O, Audouard Fericgla M, Valls J, Palomera E, Cunillera R, Palomeras E, Ibanez JM, Clave P. Healthcare costs of post-stroke oropharyngeal dysphagia and its complications: malnutrition and respiratory infections. Eur J Neurol. 2021 Nov;28(11):3670-3681. doi: 10.1111/ene.14998. Epub 2021 Jul 27. PMID 34176195
- [Background] Kim DY, Park HS, Park SW, Kim JH. The impact of dysphagia on quality of life in stroke patients. Medicine (Baltimore). 2020 Aug 21;99(34):e21795. doi: 10.1097/MD.0000000000021795. PMID 32846813
- [Background] Bath PM, Lee HS, Everton LF. Swallowing therapy for dysphagia in acute and subacute stroke. Cochrane Database Syst Rev. 2018 Oct 30;10(10):CD000323. doi: 10.1002/14651858.CD000323.pub3. PMID 30376602
- [Background] Krajczy E, Krajczy M, Luniewski J, Bogacz K, Szczegielniak J. Assessment of the effects of dysphagia therapy in patients in the early post-stroke period: a randomised controlled trial. Neurol Neurochir Pol. 2019;53(6):428-434. doi: 10.5603/PJNNS.a2019.0053. Epub 2019 Nov 14. PMID 31724147
- [Background] Sura L, Madhavan A, Carnaby G, Crary MA. Dysphagia in the elderly: management and nutritional considerations. Clin Interv Aging. 2012;7:287-98. doi: 10.2147/CIA.S23404. Epub 2012 Jul 30. PMID 22956864
- [Background] Pierpoint M, Pillay M. Post-stroke dysphagia: An exploration of initial identification and management performed by nurses and doctors. S Afr J Commun Disord. 2020 May 28;67(1):e1-e13. doi: 10.4102/sajcd.v67i1.625. PMID 32501033
- [Background] Shimizu A, Fujishima I, Maeda K, Murotani K, Ohno T, Nomoto A, Nagami S, Nagano A, Sato K, Ueshima J, Inoue T, Shimizu M, Ishida Y, Kayashita J, Suenaga M, Mori N. Delayed Dysphagia May Be Sarcopenic Dysphagia in Patients After Stroke. J Am Med Dir Assoc. 2021 Dec;22(12):2527-2533.e1. doi: 10.1016/j.jamda.2021.07.013. Epub 2021 Aug 11. PMID 34389335
- [Background] Benfield JK, Wilkinson G, Everton LF, Bath PM, England TJ. Diagnostic accuracy of the Dysphagia Trained Nurse Assessment tool in acute stroke. Eur J Neurol. 2021 Aug;28(8):2766-2774. doi: 10.1111/ene.14900. Epub 2021 May 29. PMID 33960075
- [Background] Marin S, Serra-Prat M, Ortega O, Clave P. Healthcare-related cost of oropharyngeal dysphagia and its complications pneumonia and malnutrition after stroke: a systematic review. BMJ Open. 2020 Aug 11;10(8):e031629. doi: 10.1136/bmjopen-2019-031629. PMID 32784251
- [Background] Li C, Qiu C, Shi Y, Yang T, Shao X, Zheng D. Experiences and perceptions of stroke patients living with dysphagia: A qualitative meta-synthesis. J Clin Nurs. 2022 Apr;31(7-8):820-831. doi: 10.1111/jocn.15995. Epub 2021 Aug 8. PMID 34369025
- [Background] Dziewas R, Michou E, Trapl-Grundschober M, Lal A, Arsava EM, Bath PM, Clave P, Glahn J, Hamdy S, Pownall S, Schindler A, Walshe M, Wirth R, Wright D, Verin E. European Stroke Organisation and European Society for Swallowing Disorders guideline for the diagnosis and treatment of post-stroke dysphagia. Eur Stroke J. 2021 Sep;6(3):LXXXIX-CXV. doi: 10.1177/23969873211039721. Epub 2021 Oct 13. PMID 34746431
- [Background] Jones CA, Colletti CM, Ding MC. Post-stroke Dysphagia: Recent Insights and Unanswered Questions. Curr Neurol Neurosci Rep. 2020 Nov 2;20(12):61. doi: 10.1007/s11910-020-01081-z. PMID 33136216
- [Background] Fang WJ, Zheng F, Zhang LZ, Wang WH, Yu CC, Shao J, Wu YJ. Research progress of clinical intervention and nursing for patients with post-stroke dysphagia. Neurol Sci. 2022 Oct;43(10):5875-5884. doi: 10.1007/s10072-022-06191-9. Epub 2022 Jun 4. PMID 35661279
- [Background] King D, Wittenberg R, Patel A, Quayyum Z, Berdunov V, Knapp M. The future incidence, prevalence and costs of stroke in the UK. Age Ageing. 2020 Feb 27;49(2):277-282. doi: 10.1093/ageing/afz163. PMID 31957781

DOCUMENTS (2):
  • Statistical Analysis Plan (2026-01-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT07267468/SAP_000.pdf
  • Informed Consent Form (2025-10-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT07267468/ICF_001.pdf